CLINICAL TRIAL: NCT00674505
Title: FiberNet Renal Artery Embolic Protection Study: A Prospective, Single-arm Feasibility Trial of Renal Artery Distal Protection Using the Lumen Biomedical FiberNet Embolic Protection System
Brief Title: Safety & Performance Study of Lumen Biomedical's FiberNet Distal Protection System for the Treatment of Renal Artery Stenosis
Acronym: FORTRESS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: VIVA Physicians (Other)
Collaborators: Lumen Biomedical (Industry); Prairie Education and Research Cooperative (Industry)
Responsible Party: John R. Laird, MD, University of California, Davis
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: G070189/S002
Record Dates: First submitted 2008-05-06; First posted 2008-05-08 (Estimated); Last update posted 2010-02-17 (Estimated); Status verified 2010-02

CONDITIONS: Renal Stenting in the Treatment of Pts w/a High Grade Ostial Atherosclerotic Renal Lesion(s).

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment, Open label, Single Group Assignment (Other)
  Interventions: Device: Lumen Biomedical FiberNet Embolic Protection System

INTERVENTIONS:
Device: Lumen Biomedical FiberNet Embolic Protection System — to demonstrate the safety and filter efficiency of the Lumen Biomedical FiberNet Embolic Protection System during the performance of primary renal stenting in the treatment of pts with a high grade ostial atherosclerotic renal lesion(s).

SUMMARY:
To evaluate the procedural safety and filter efficiency of the FiberNet® Embolic Protection System when used in conjunction with the Boston Scientific Express SD Stent System for primary stenting of ostial atherosclerotic renal lesions in patients with atherosclerotic renal artery stenosis.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 and ≤ 85 years.
2. Subject or subject's legal representative have been informed of the nature of the study, agrees to participate and has signed an IRB approved consent form.
3. Subject understands the duration of the study and it's follow up visit requirements.
4. Unilateral or bilateral atherosclerotic de novo renal artery stenosis (RAS) associated with any or all of the following:

   1. SBP >140 despite ≥3 anti-hypertensive medications
   2. Estimated Glomerular Filtration Rate (eGFR) ≥30-≤70 cc/min calculated using the Modified Diet in Renal Disease (MDRD) formula
   3. Recurrent episodes of decompensated heart failure
   4. Recurrent episodes of "flash" pulmonary edema

Angiographic Inclusion Criteria

1. ≥70% <100% renal artery stenosis (by visual estimate) involving unilateral, bilateral renal arteries or solitary renal artery.
2. Renal pole-to-pole length >7cm.
3. Lesion ≤15 mm from the aorto-ostial junction.
4. Renal artery reference lumen diameter ≥3.5 - ≤7 mm for FiberNet placement.

Exclusion Criteria:

Clinical Exclusion Criteria

1. Estimated life expectancy <12 months.
2. Estimated Glomerular Filtration Rate (eGFR) <30 cc/min.
3. Renal pole-to-pole length <7cm on side of diseased kidney.
4. No history of transplanted kidneys or polycystic kidney disease.
5. Uncontrolled hypercoagulability.
6. Known allergies or sensitivities to heparin, aspirin, other anti-coagulant/antiplatelet therapies, nitinol and stainless steel.
7. Known allergy to contrast media that cannot adequately be pre-medicated prior to study procedure.
8. Patient refuses possible temporary or permanent hemodialysis.
9. Refuses possible surgery for repair of access site or renal artery.
10. Known severe coronary or carotid disease likely to require surgical treatment after enrollment or during follow-up period.
11. Uncompensated congestive heart failure.
12. Current enrollment in any investigational study wherein patient participation has not been completed.
13. Cardiovascular surgical or cardiovascular interventional procedures (including, but not limited to, aortic, renal, cardiac, carotid, femoro-popliteal, and below the knee) within 30 days prior to enrollment in this study.
14. Planned or predicted cardiovascular surgical or interventional procedures outside of the affected renal artery (including, but not limited to, aortic, renal, cardiac, carotid, contralateral femoro-popliteal, and contralateral below the knee) within 30 days after entry into this study and prior to completion of the 30 day follow-up.
15. Pregnancy, breast-feeding or plans to become pregnant in female of child bearing potential.
16. Any patient who in the opinion of the investigator would not be a good candidate for enrollment.

Angiographic Exclusion Criteria

1. Early bifurcation of the main renal artery preventing complete embolic protection of the kidney with the FiberNet.
2. Fibromuscular Dysplasia.
3. Presence of thrombus at the lesion site.
4. Non-ostial atherosclerosis (lesion >15mm from the renal ostium).
5. Subintimal guidewire placement resulting in dissection of the renal artery or aorta, or perforation of the renal artery or aorta prior to deployment of the device.
6. Severe calcification likely to prevent the passage of the device. -

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2008-01; Primary Completion 2009-06 (Estimated)

PRIMARY OUTCOMES:
Measurable amount of macro/micro atheroma particle captured by the FiberNet EPS as adjudicated by core lab analysis. | Various secondary endpoints evaluated at 30 days and 6 months

SECONDARY OUTCOMES:
Progression to temporary/permanent renal replacement therapy and Analysis of debris captured by the FiberNet® Embolic Protection System | most at 30 days and 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- VIVA Physicians Inc., San Jose, California, United States

REFERENCES:
- [Derived] Laird JR, Tehrani F, Soukas P, Joye JD, Ansel GM, Rocha-Singh K. Feasibility of FiberNet(R) embolic protection system in patients undergoing angioplasty for atherosclerotic renal artery stenosis. Catheter Cardiovasc Interv. 2012 Feb 15;79(3):430-6. doi: 10.1002/ccd.23292. Epub 2011 Dec 8. PMID 21805607